CLINICAL TRIAL: NCT04596774
Title: The Impact of Using Enhanced Recovery After Surgery Approach on Orthognathic Surgery Outcome: A Historical Cohort Study
Brief Title: The Impact of Enhanced Recovery After Surgery in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, MD, Attending Anesthesiologist, Associate Professor, Istanbul University
Other Study IDs: 2020/965
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Enhanced Recovery After Surgery; Hospital Stay; Postoperative Nausea and Vomiting; Pain, Postoperative
Keywords: Orthognathic surgery; Enhanced recovery after surgery (ERAS); Analgesia; Postoperative nausea vomiting (PONV); Satisfaction
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative; Agnosia; Personal Satisfaction | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 patients were applied traditional approach. Patients received intraoperative 10 mL/kg/h IV izolen infusion. Opioids and PONV prophylaxis were applied when required.
  Interventions: Procedure: Traditional Approach
- Group 2: Group 2 received Enhanced Recovery After Surgery (ERAS) approach. Patients did not preoperatively smoke for 48 hours, drank clear liquids until the last 2 hours and received 6 mL/kg/h IV izolen infusion intraoperatively. In these; gastric aspiration was applied before extubation, PONV prophylaxis was supported routinely, and patient controlled analgesia was added to the routine analgesia plan for the first postoperative 48 hours.
  Interventions: Procedure: Enhanced Recovery After Surgery (ERAS) Approach

INTERVENTIONS:
Procedure: Traditional Approach — Patients received intraoperative 10 mL/kg/h IV izolen infusion. Opioids and PONV prophylaxis were applied when required.
  Groups: Group 1
Procedure: Enhanced Recovery After Surgery (ERAS) Approach — Patients did not preoperatively smoke for 48 hours, drank clear liquids until the last 2 hours and received 6 mL/kg/h IV izolen infusion intraoperatively. In these; gastric aspiration was applied before extubation, PONV prophylaxis was supported routinely, and patient controlled analgesia was added to the routine analgesia plan for the first postoperative 48 hours.
  Groups: Group 2

SUMMARY:
Aim: Orthognathic surgeries are generally associated with blood loss, swelling, postoperative nausea vomiting (PONV), and pain. The aim of this study is to improve postoperative outcome in patients undergoing orthognatic surgeries by the use of Enhanced Recovery After Surgery (ERAS) protocols.

Material methods: After Ethics Committee approval (2020/965), the data of 90 patients who underwent elective orthognathic surgery, were investigated. Following standard monitorization and general anesthesia; Group 1 patients were applied traditional approach and received intraoperative 10 mL/kg/h IV izolen infusion. Group 2 received ERAS approach. Patients in Group 2 did not preoperatively smoke for 48 hours, drank clear liquids until the last 2 hours, and received 6 mL/kg/h IV izolen intraoperatively. In these; gastric aspiration was also applied before extubation, PONV prophylaxis and patient controlled analgesia was added to the routine plans for the first postoperative 48 hours. The primary endpoint was length of hospital stay. The secondary endpoints were intraoperative follow-up data, length of postanesthesia care unit (PACU) stay, numeric rating scale (NRS) pain scores, opioid consumption and PONV incidences through the postoperative first 48 hours, and satisfaction scores.

DETAILED DESCRIPTION:
Aim: Orthognathic surgeries are extensive surgeries including both soft and hard tissues of the facial region of the skull associated with blood loss, inflammatory reactions, massive swelling, postoperative nausea vomiting (PONV), and severe pain. Therefore; in most of the patients who are with dentofacial deformity and undergo orthognathic surgery, postoperative recovery generally requires a long troublesome period. The aim of this study is to improve postoperative outcome by the use of Enhanced Recovery After Surgery (ERAS) protocols.

Material methods: After Ethics Committee approval (2020/965), the data of 90 patients who underwent elective orthognathic surgery, were investigated. Following standard monitorization and general anesthesia; Group 1 patients were applied traditional approach and received intraoperative 10 mL/kg/h IV izolen infusion. Rescue analgesics and PONV prophylaxis were applied when required through the postoperative first 48 hours. Group 2 received ERAS approach. Patients in Group 2 did not preoperatively smoke for 48 hours, drank clear liquids until the last 2 hours, and received 6 mL/kg/h IV izolen infusion intraoperatively. In these; gastric aspiration was also applied before extubation, PONV prophylaxis was supported routinely, and patient controlled analgesia was added to the routine analgesia plan for the first postoperative 48 hours. The primary endpoint was length of hospital stay. The secondary endpoints were intraoperative follow-up data, numeric rating scale (NRS) pain scores, opioid consumption, PONV incidences, length of postanesthesia care unit (PACU) stay, satisfaction scores of two groups through the postoperative first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthognathic surgery (bimaxillary, mandibular/maxillary)
* Patients aged between 18 and 40 years of age
* American Society of Anesthesiologists (ASA) physical status of 1-2
* Capable of understanding the instructions for using the NRS pain scores
* Capable of replying the study-based questions
* Absence of mental/psychiatric disorders
* Absence of chronic analgesic/opioid use
* Absence of alcohol/illicit drug use

Exclusion Criteria

* Patients who are younger than 18 years of age
* Patients who are older than 45 years of age
* American Society of Anesthesiologists (ASA) physical status of 3-4
* Not capable of consenting
* Not capable of understanding the instructions for using the NRS pain
* scores
* Not capable of replying the study-based questions
* Presence of mental/psychiatric disorders
* Presence of chronic analgesic/opioid use
* Presence of alcohol/illicit drug use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients eligible for orthognathic surgery Patients who were operated under either the traditional approach or the Enhanced Recovery After Surgery (ERAS) approach Patients aged between 18 and 40 years of age American Society of Anesthesiologists (ASA) physical status of 1-2
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 0-48 hours
  Post Anaesthetic Discharge Scoring System (PADSS) (≥9/10)

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | 0-5 hours
  Intraoperative follow-up
Heart rate | 0-5 hours
  Intraoperative follow-up
Intraoperative fentanyl requirement | 0-5 hours
  Intraoperative follow-up
The amount of blood loss | 0-5 hours
  Intraoperative follow-up (aspirator and gases)
The difference of preoperative-postoperative haemoglobin values | 0-12 hours
  Preop Hb-Postop Hb
Length of stay in postoanesthesia care unit (PACU) | 0-1 hours
  Modified Aldrete Scoring system (≥9/10)
Pain (Numeric rating scale (NRS)) scores | 0-48 hours
  Postoperative Numeric rating scale (NRS) pain scores (0: no pain, 10: worst pain imaginable)
Opioid (meperidine) consumption | 0-48 hours
  Amount of opioid administered to the patient through the postoperative first 48 hours (Group 1: NRS≥4, Group 2: Patient controlled analgesia system)
Incidence of postoperative nausea and vomiting (PONV) | 0-48 hours
  Number of feeling nausea or vomiting (on postoperative days 1 and 2)
Postoperative first oral intake | 0-24 hours
  First oral liquid (water) intake time (postoperatively as soon as possible)
Postoperative first passage of flatus or stool | 0-24 hours
  First passage of flatus or stool (postoperatively as soon as possible)
Postoperative first mobilization | 0-24 hours
  First mobilization time (standing up-walking for any reason) (postoperatively as soon as possible)
Patient satisfaction | 0-48 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied
Surgeon satisfaction | 0-48 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, MD,AssocProf, Principal Investigator — Study Principal Investigator, Corresponding author
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dobbeleir M, De Coster J, Coucke W, Politis C. Postoperative nausea and vomiting after oral and maxillofacial surgery: a prospective study. Int J Oral Maxillofac Surg. 2018 Jun;47(6):721-725. doi: 10.1016/j.ijom.2017.11.018. Epub 2018 Jan 1. PMID 29301675
- [Result] Lin S, McKenna SJ, Yao CF, Chen YR, Chen C. Effects of Hypotensive Anesthesia on Reducing Intraoperative Blood Loss, Duration of Operation, and Quality of Surgical Field During Orthognathic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2017 Jan;75(1):73-86. doi: 10.1016/j.joms.2016.07.012. Epub 2016 Jul 25. PMID 27542543
- [Result] Mobini A, Mehra P, Chigurupati R. Postoperative Pain and Opioid Analgesic Requirements After Orthognathic Surgery. J Oral Maxillofac Surg. 2018 Nov;76(11):2285-2295. doi: 10.1016/j.joms.2018.05.014. Epub 2018 May 19. PMID 29886112
- [Result] Agbaje J, Luyten J, Politis C. Pain Complaints in Patients Undergoing Orthognathic Surgery. Pain Res Manag. 2018 Jul 15;2018:4235025. doi: 10.1155/2018/4235025. eCollection 2018. PMID 30123397